CLINICAL TRIAL: NCT02876627
Title: The Effect of 12 Weeks of Aerobic Training Program on Erythrocyte Levels in Women With Breast Cancer After Chemotherapy
Brief Title: Effect Aerobic Training on Women With Breast Cancer After Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Isfahan (Other)
Responsible Party: Principal Investigator, Prof.Mehdi Kargarfard, Principal Investigator, University of Isfahan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201527904IR
Record Dates: First submitted 2016-08-15; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Cancer; Exercise; Hemoglobins
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

ARMS (1):
- breast cancer (Experimental): Effect of exercise training on breast cancer patient
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — twelve-week aerobic exercise training program consisted of three sessions per week, each session lasting 30 to 60 minutes 50 to 75 percent of their maximum heart rate reserve

SUMMARY:
Introduction: The purpose of this study was to determine the effect of twelve weeks of aerobic exercise program on erythrocyte levels in women with breast cancer after chemotherapy.

Methods: Thirty women with breast cancer after chemotherapy of Sydalshhda hospital (aged between 47-65 years) volunteered for this study, and then randomly selected an exercise (n = 15) and control (n = 15) groups. Exercise group completed a twelve-week aerobic exercise training program consisted of three sessions per week, each session lasting 30 to 60 minutes 50 to 75 percent of their maximum heart rate reserve, while the control group were followed. Blood samples including red blood cell counts (RBC), hematocrit (HCT), hemoglobin (HB), peak oxygen consumption before and after 12 weeks of aerobic exercise were measured. For analysis of data, repeated-measures analysis of variance (ANOVA) was used.

ELIGIBILITY:
Inclusion Criteria:

women with breast cancer , who can do a physical, physiological and psychological test; and did not have exercise limitations due to neuromuscular and/or musculoskeletal disease; did not have any health problems that prevented maximum effort on the treadmill test.

Exclusion Criteria:

women under erythropoietin treatments, uncontrolled cardiovascular or pulmonary diseases, uncontrolled arrhythmias, orthopedic conditions that would limit exercise participation, refusal for randomization, or participation in aerobic exercise training within 3 months before beginning the study.

Ages: 47 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
effect of exercise on CBC parameters (measured by ELISA methods) | up to 12 weeks

SECONDARY OUTCOMES:
effect of exercise on peak oxygen consumption, measured by vo2 max test | up to 12 weeks